CLINICAL TRIAL: NCT02501785
Title: Caregiver Burden Within the Ambulatory Extended Recovery (AXR) Patient Population
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-145
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Caregiver Burden
Keywords: Quality of Life; Patient care givers; 15-145; Ambulatory Extended Recovery
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patient and caregivers: This is a prospective cohort study. Four questionnaires will be used to collect data from caregivers: demographic and socioeconomic data will be collected from the caregiver before the patient's surgery, and caregiver burden information will be collected 15 (+/- 3) days after surgery.
  Interventions: Behavioral: Caregiver Reaction Assessment (CRA); Behavioral: The Caregiver Quality of Life - Cancer (CQOLC)

INTERVENTIONS:
Behavioral: Caregiver Reaction Assessment (CRA)
Behavioral: The Caregiver Quality of Life - Cancer (CQOLC)

SUMMARY:
The purpose of this study is to understand the level of caregiver burden related to caring for a patient who goes home within the first 24 hours following surgery. As the caregiver they are providing care to a family member, friend, or neighbor. Even when not formally trained, the care they provide is important to the patient's recovery. Providing care in this manner can be stressful. This study will help us understand what aspects of the patient's recovery are most difficult for the caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver/patient pairs undergoing surgery for an indication tracked within the Breast, Gynecology, Head and Neck, and Urology AXR program
* English speaking
* Patients willing to provide demographic, surgical, and outcome information
* Caregivers willing to provide demographic, socioeconomic, and caregiver experience information
* Caregivers willing to complete the caregiver burden measurement scales

Exclusion Criteria:

* Patients undergoing surgery within the AXR pathway that do not have a caregiver
* Non-English speaking patients or caregivers
* Patients unwilling to provide demographic and surgical information
* Caregivers unwilling to provide demographic, socioeconomic, or caregiver experience information or unwilling to complete the caregiver burden measurement scales

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and caregivers will be recruited prior to the patient's scheduled surgery during a clinic visit within the four target services. (Breast, Gynecology, Head and Neck, and Urology
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Caregiver Reaction Assessment (CRA) score | 1 year
  in the AXR patient population. Burden will be defined as both a total CRA score and sub scores and will be summarized using descriptive statistics. CRA total score of 72 and subscale scores of 3 or greater will be used to indicate high levels of caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Sovel, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/